CLINICAL TRIAL: NCT06086483
Title: Pain Management and Functional Recovery After Adductor Canal Block Combined With iPACK Block for Total Knee Arthroplasty. A Prospective, Randomized, Double-blinded Clinical Trial.
Brief Title: Pain Management After Adductor Canal Block for Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 495/2020
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis; Knee Arthritis; Knee Arthropathy; Knee Pain Chronic
Keywords: iPACK; Adductor Canal Block; pain management; multimodal analgesia; peripheral nerve block; knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia | interventions — Ropivacaine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPACK block+ABC block (Active Comparator): Patients received a preoperative ultrasound-guided iPACK block with 20 mL of 0.25% ropivacaine and an Adductor Canal block with 20mL 0.25% ropivacaine.
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- Sham blocks (Active Comparator): Patients received a preoperative ultrasound-guided iPACK block with 20 mL of 0.9% normal saline and an Adductor Canal block with 20mL 0.9% normal saline.
  Interventions: Drug: 0.9%sodium chloride

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution — 20 mL 0.5% ropivacaine was injected into the PENG block
  20 mL 0.5% ropivacaine was injected into the Adductor Canal block
  Other Names: Ropimol
  Arms: iPACK block+ABC block
Drug: 0.9%sodium chloride — 20 mL 0.9% sodium chloride was injected into the PENG block
  20 mL 0.5% sodium chloride was injected into the Adductor Canal block
  Other Names: normal saline
  Arms: Sham blocks

SUMMARY:
This randomized, double-blinded, placebo-controlled trial sought to evaluate the efficacy of the iPACK block with Adductor Canal Block on postoperative pain, functional recovery and NLR and PLR levels.

DETAILED DESCRIPTION:
The Interspace between the popliteal artery and capsule of the posterior knee, or iPACK block, together with the Adductor Canal block (ACB), has been described and shows promise in providing analgesia to the knee joint. However, the effect of these two blocks on postoperative pain levels, functional recovery, and stress response is uncertain. This study compares a preoperative iPACK and ACB block to Sham blocks before total knee arthroplasty under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old undergoing unilateral total knee arthroplasty

Exclusion Criteria:

* refusal to participate
* < 18 yo
* Chronic opioid use
* localized infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
postoperative Numeric Pain Rating Scale | 24 hours after surgery
  Numeric Pain Rating Scale. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
postoperative Numeric Pain Rating Scale et rest | 48 hours after surgery
  Numeric Pain Rating Scale. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
postoperative Numeric Pain Rating Scale et rest | 72 hours after surgery
  Numeric Pain Rating Scale. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
postoperative Numeric Pain Rating Scale et rest | 96 hours after surgery
  Numeric Pain Rating Scale. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
postoperative Numeric Pain Rating Scale during active flexion | 48 hours after surgery
  Numeric Pain Rating Scale. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
postoperative Numeric Pain Rating Scale during active flexion | 72 hours after surgery
  Numeric Pain Rating Scale. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
postoperative Numeric Pain Rating Scale during active flexion | 96 hours after surgery
  Numeric Pain Rating Scale. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")

SECONDARY OUTCOMES:
Postoperative opioid consumption | 96 hours after surgery
  milligrams of intravenous morphine equivalents
Neutrophil-to-lymphocyte ratio | 12 hours after surgery
  Neutrophil-to-lymphocyte ratio
Neutrophil-to-lymphocyte ratio | 24 hours after surgery
  Neutrophil-to-lymphocyte ratio
Platelet-to-lymphocyte ratio | 12 hours after surgery
  Platelet-to-lymphocyte ratio
Platelet-to-lymphocyte ratio | 24 hours after surgery
  Platelet-to-lymphocyte ratio
Time to first opioid administration | 96 hours postoperatively
  Hours to first administration of an intravenous opioid drug

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Żaba, Ph.D., Study Chair — Department of Emergency Medicine Clinic; Malgorzata Domagalska, Ph.D., Principal Investigator — Department of Palliative Medicine, University of Medical Sciences, Poznań, Poland
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: Yes
The data presented in this study are available on request from the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December 2024
Access Criteria: The data presented in this study are available on request from the corresponding author.